CLINICAL TRIAL: NCT05251012
Title: Three-dimensional Quantitative Flow Ratio (3D-QFR) in Non-selected Angiographic Stenosis. A Spanish Multicentre Study.
Brief Title: 3D-QFR in Non-selected Angiographic Stenosis. A Spanish Multicentre Study.
Status: Completed | Type: Observational
Sponsor: Pablo Manuel Fernandez Corredoira (Other)
Collaborators: Hospital Clínico Universitario Lozano Blesa (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Hospital General de Ciudad Real (Other); Hospital de Leon (Other Government); Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Sponsor-Investigator, Pablo Manuel Fernandez Corredoira, Cardiology resident, Hospital Miguel Servet
Organization: Hospital Miguel Servet (Other)
Other Study IDs: 1.1
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Coronary Stenosis; Coronary Artery Disease
Keywords: Quantitative Flow Ratio; Coronary physiology; Computational physiology
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Physiology-based decision-making about the need for revascularisation in patients with stable coronary heart disease has consistently proven better clinical outcomes than a merely anatomical approach. However, against the current recommendations, revascularisation in most of patients with chronic coronary syndromes still relies on coronary angiography alone. The increase in costs and in procedural complexity of wire-based physiology may explain the latter. Therefore, a novel non-invasive functional quantitative flow ratio (QFR) index was created in order to solve it.

A retrospective and multicentre study is performed to assess the 5-year prognosis of patients undergoing coronary angiography through a centralized QFR analysis. Consecutive participants with confirmed or suspected diagnosis of stable coronary disease who underwent a coronary angiography between 01/01/2015 and 12/31/2015 were included.

Aims of the study:

* To evaluate the prognosis of stable coronary disease depending on the functional assessment of coronary artery disease.
* To determine the % of percutaneous coronary interventions that could be avoided if this study had been carried out through functional assessment of coronary artery disease based on 3-dimensional vessel reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive participants with confirmed or suspected diagnosis of stable coronary disease who underwent a coronary angiography between 01/01/2015 and 12/31/2015.

Exclusion Criteria:

1. Previous coronary artery bypass grafting.
2. <18 years or >90 years.
3. Angiographic acquisitions that make it impracticable to perform QFR analysis (patients will be included for descriptive purposes).
4. If a patient has undergone several unscheduled coronary angiographies during the study period, the first will be included as the index case and the following as a follow-up event.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive participants with confirmed or suspected diagnosis of stable coronary disease who underwent a coronary angiography between 01/01/2015 and 12/31/2015.
Sampling Method: Non-Probability Sample
Enrollment: 803 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
To assess the 5-year prognosis of patients undergoing coronary angiography with confirmed or suspected diagnosis of stable coronary disease. | 5 years.
To define the functional index of revascularized and non-revascularized coronary stenosis and to analyse the prognosis according to the result and the treatment performed. | 5 years.
To determine number of percutaneous coronary intervention procedures performed on non-significant stenosis through QFR analysis and their prognosis. | 5 years.
To evaluate the prognosis of non-revascularized and functionally significant coronary artery disease using QFR. | 5 years.